CLINICAL TRIAL: NCT04141241
Title: Multi-center, Randomized, Double-blinded, Placebo-controlled, Parallel-design, 12-week, Therapeutic Exploratory, Phase 2a Study to Evaluate the Safety and Efficacy of PH100 Tablet in T2DM Patients With Recent Cardiovascular Complications
Brief Title: Phase 2a Study to Evaluate the Safety and Efficacy of PH100 Tablet in T2DM Patients With Recent Cardiovascular
Acronym: PH100_IIa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bota Bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BOTAB-DBCVC-PH100
Record Dates: First submitted 2019-10-21; First posted 2019-10-28 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Type 2 Diabetes Mellitus With Circulatory Complciation
Keywords: T2DM with Recent Cardiovascular Complications

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose PH100: 800mg/day (Experimental): * PH100 (Ecklonia cava Phlorotannin) 200mg/tablet
  * PH100 2 tablets (400mg) and Placebo 2 tablets BID during 12wks
  Interventions: Drug: Ecklonia cava Phlorotannin
- High Dose PH100: 1600mg/day (Experimental): - PH100 4 tablets (800mg) BID during 12wks
  Interventions: Drug: Ecklonia cava Phlorotannin
- Placebo (Placebo Comparator): * Placebo 200mg/tablet
  * Placebo 4 tablets BID during 12wks
  Interventions: Drug: Ecklonia cava Phlorotannin

INTERVENTIONS:
Drug: Ecklonia cava Phlorotannin — Drugs that have been administered prior to participation in this study that are not expected to affect the results of this study will be accepted at the investigator's discretion.
  Other Names: PH100

SUMMARY:
This is a Multi-center, Randomized, Double-blinded, Placebo-controlled, Parallel-design, 12-Week, Therapeutic exploratory, Phase IIa Study which will patients with type 2 diabetes mellitus and recent cardiovascular complications.

DETAILED DESCRIPTION:
After a screening, 114 patients will be stratified randomized in a 1:1:1 ratio to the 3 arms (PH100 800mg/day, PH100 1600mg/day, Placebo) to evaluate the safety and efficacy of PH100.

Subjects will visit the centers on Week 4, 8 and 12 during the entire 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 19 years old
2. Subjects who have been treated for cardiovascular complications (stent insertion due to angina pectoris, myocardial infarction, cerebral ischemia, peripheral vascular disease) within 4 weeks prior to baseline
3. T2DM patients who diagnosed with type 2 diabetes prior to or above cardiovascular complications and have been taking oral hypoglycemic agents and/or receiving insulin treatment before the above complication occurred
4. Subjects taking a stable dose of statins and are anticipated to have no change in dose during the duration of the study
5. The following is confirmed through screening:

   * AST/ALT ≤ 2.5 X ULN
   * Creatinine ≤ 1.5 X ULN
   * Hemoglobin ≥ 10 g/dL
   * 6.5% ≤ HbA1c ≤ 11%
6. Women of child-bearing potential who have negative pregnancy testing results and have agreed to use appropriate measures of contraception* during the duration of the study (*appropriate contraception is defined as women of child-bearing potential, excluding women in whom more than 52 weeks have passed since their last period, using the following methods: surgical sterilization, intrauterine device, condoms, barrier contraceptives, absolute abstinence)
7. Subjects who have signed the informed consent form (or whose legal representative has signed) and who are deemed to be able to follow the requirements of the study

Exclusion Criteria:

1. T2DM patients, secondary DM patients, Gestational DM patients
2. Subjects who have a history of secondary hypertension or have a disease history of suspicious secondary hypertension. This includes but is not restricted to: aortic coarctation, primary hyperaldosteronism, renal artery stenosis, Cushing's disease, pheochromocytoma, polycystic kidney disease, etc.
3. Subjects taking anti-inflammatory agents including corticosteroids/NSAIDs (However, maximum 100mg of aspirin per day is allowed)
4. Subjects with chronic liver/renal disease or malignancy
5. Supplements containing kajime or kajime derivatives (e.g. Seapolynol, Fibroboost, Fibronol, Seanol Longevity Plus, Circulate, Alginol, PC Eckonia Cava, Seanol, Seanol-F, Seanol-EX, Seanol-TX, Venusen, Memories with Seanol-P, Astaxanthol, Brilliant Vision with Seanol-P, Gly-Control, Gyne-Andro-Plex, Lipid Balance, Seanol with Broccoraphanin, Marine D3, Botabio everyone, Botabio power, Botabio red, Botabio premium, Botabio Eplus) and related medications, or subjects who have a history of hypersensitivity to high iodine containing products (seaweed, shellfish, etc.)
6. Pregnant, breast-feeding subjects or subjects who have plans for pregnancy
7. Subjects who have taken supplements containing kajime or kajime derivatives within 4 weeks of baseline (e.g., Seapolynol, Fibroboost, Fibronol, Seanol Longevity Plus, Circulate, Alginol, PC Eckonia Cava, Seanol, Seanol-F, Seanol- EX, Seanol-TX, Venusen, Memories with Seanol-P, Astaxanthol, Brilliant Vision with Seanol-P, Gly-Control, Gyne-Andro-Plex, Lipid Balance, Seanol with Broccoraphanin, Marine D3, Botabio everyone, Botabio power, Botabio red, Botabio premium, Botabio Eplus)
8. Subjects who have participated in another clinical trial within 4 weeks of baseline and have taken other clinical trial medications
9. Subjects who have received treatment for or who test positive for HBsAg, HCV antibody, or HIV at baseline
10. Subjects who have an acute inflammatory disease other than cardiovascular complications within 4 weeks of baseline
11. Subjects who have gastrointestinal diseases that may affect the absorption, distribution, metabolism, and excretion of drugs (e.g. Crohn's disease) and subjects who have a history of gastrointestinal surgery (with the exception of appendectomy and hernia repair), or subjects with active gastritis, gastrointestinal/rectal bleeding, active inflammatory bowel disease within the past 12 months
12. Subjects with autoimmune disease (e.g. rheumatoid arthritis) or who require chronic anti-inflammatory treatment
13. Subjects with a history of drug or alcohol abuse
14. Subjects who are judged not to be appropriate for participation in the study or who have a medical condition that may have an influence on the study results

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
hs-CRP (high-sensitivity C-reactive protein) | Visit 2(Baseline Visit) vs Visit 5(week 12)
  Change in hs-CRP level compared to baseline after 12 weeks of investigational product administration

SECONDARY OUTCOMES:
hs-CRP | Visit 2(Baseline Visit), Visit 3(week 4), Visit 4(week 8)
  Change in hs-CRP level compared to baseline after 4 weeks, 8 weeks of investigational product administration
hs-CRP: monthly rate of change | Between Visit 2(Baseline Visit) and Visit 3(week 4), Between Visit 3(week 4) and Visit 4(week 8), Between Visit 4(week 8) and Visit 5(week 12)
  Change in hs-CRP level monthly
Interleukin-6 (IL-6) | Visit 2(Baseline Visit), Visit 3(week 4), Visit 4(week 8), Visit 5(week 12)
  Change in IL-6 [Inflammatory Marker]
Tumor Necrosis Factor-α (TNF- α) | Visit 2(Baseline Visit), Visit 3(week 4), Visit 4(week 8), Visit 5(week 12)
  Change in TNF- α [Inflammatory Marker]
Malondialdehyde (MDA) | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in MDA [Biomarkers of oxidative stress]
Oxidized Low Density Lipoprotein (Oxidized LDL) | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in Oxidized LDL [Biomarkers of oxidative stress]
Glutathione Peroxidase (GPX) | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in GPX [Biomarkers of oxidative stress]
Superoxide Dismutase (SOD) | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in SOD [Biomarkers of oxidative stress]
Total AntiOxidants (TAS) | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in TAS [Biomarkers of oxidative stress]
HbA1c | Visit1(screening), Visit 5(week 12)
  Change in HbA1c level compared to Visit1(screening) after 12 weeks of investigational product administration
Adiponectin | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in Adiponectin level compared to Visit 2(Baseline Visit) after 12 weeks of investigational product administration
Free Fatty Acid | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in Free Fatty Acid level compared to Visit 2(Baseline Visit) after 12 weeks of investigational product administration
High Density Lipoprotein-cholesterol (HDL-C) | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in HDL-C level compared to Visit 2(Baseline Visit) after 12 weeks of investigational product administration [Lipid Profile]
Low Density Lipoprotein-cholesterol (LDL-C) | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in LDL-C level compared to Visit 2(Baseline Visit) after 12 weeks of investigational product administration [Lipid Profile]
Triglyceride (TG) | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in TG level compared to Visit 2(Baseline Visit) after 12 weeks of investigational product administration [Lipid Profile]
Total Cholesterol (TC) | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in TC level compared to Visit 2(Baseline Visit) after 12 weeks of investigational product administration [Lipid Profile]
Homocysteine | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in Homocysteine level compared to Visit 2(Baseline Visit) after 12 weeks of investigational product administration
Fibrinogen | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in Fibrinogen level compared to Visit 2(Baseline Visit) after 12 weeks of investigational product administration
MACE (Major Adverse Cardiovascular Events) | Visit 3(week 4), Visit 4(week 8), Visit 5(week 12)
  Incidence rate of MACE (Major Adverse Cardiovascular Events) during investigational product administration
Left Ventricular Ejection Fraction | Visit 2(Baseline Visit), Visit 5(week 12)
  Change in LVEFF compared to Visit 2(Baseline Visit) after 12 weeks of investigational product administration by Echocardiogram
Blood Pressure (Systolic Blood Pressure, Diastolic Blood Pressure) | Visit 2(Baseline Visit), Visit 3(week 4), Visit 4(week 8), Visit 5(week 12)
  Change in SiSBP, SiDBP
BMI | Visit 2(Baseline Visit), Visit 3(week 4), Visit 4(week 8), Visit 5(week 12)
  Change in BMI
Waist-hip ratio | Visit 2(Baseline Visit), Visit 3(week 4), Visit 4(week 8), Visit 5(week 12)
  Change in Waist-hip ratio
AE (Adverse Events) | Visit 2(Baseline Visit), Visit 3(week 4), Visit 4(week 8), Visit 5(week 12)
  [Safety and Tolerability] Incidence of AEs during investigational product administration
Pulse | Visit 1(Screening), Visit 2(Baseline Visit), Visit 3(week 4), Visit 4(week 8), Visit 5(week 12)
  [Safety and Tolerability] Check the Vital Sign (pulse) every visit schedule
Body Temperature | Visit 1(Screening), Visit 2(Baseline Visit), Visit 3(week 4), Visit 4(week 8), Visit 5(week 12)
  [Safety and Tolerability] Check the Vital Sign (body temperature) every visit schedule

IPD SHARING:
Plan to Share IPD: No